CLINICAL TRIAL: NCT00599950
Title: Anterior Stromal Changes After PRK by Using Intraoperative Mitomicin C.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Asociación para Evitar la Ceguera en México, Asociación para Evitar la Ceguera en México
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cornea 4
Record Dates: First submitted 2008-01-08; First posted 2008-01-24 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Refractive Disorders
Keywords: Mitomycin C; Corneal epithelium; Photorefractive keratectomy (PRK); Confocal microscope
MeSH Terms: conditions — Refractive Errors | interventions — Mitomycin; Photorefractive Keratectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Topical mitomycin C on the corneal epithelium of patients undergoing photorefractive keratectomy (PRK)
  Interventions: Drug: Mitomycin C and Photorefractive keratectomy (PRK)
- 2 (Placebo Comparator): Photorefractive keratectomy (PRK)without mitomycin C.
  Interventions: Drug: Mitomycin C and Photorefractive keratectomy (PRK)

INTERVENTIONS:
Drug: Mitomycin C and Photorefractive keratectomy (PRK) — Topical mitomycin C on the corneal epithelium of patients undergoing photorefractive keratectomy (PRK)

SUMMARY:
To evaluate the confocal microscopy changes in keratocyte density at the anterior stromal after Photorefractive keratectomy (PRK) surgery, using intraoperative mitomycin C(Mitolem, LEMERY, S.A. de C.V. Mexico D.F. Reg. 136M92 SSA).

DETAILED DESCRIPTION:
10 eyes of 10 patients underwent PRK,using intraoperative mitomycin C (Mitolem, LEMERY, S.A. de C.V. Mexico D.F. Reg. 136M92 SSA), and 10 eyes for the same patients underwent PRK without intraoperative mitomycin C. A central scan of the total corneal thickness was taken with the confocal microscope (Confoscan 4, Fortune Technologies, Italy) after surgery, and 1 week, 1 month, 3 months, and 6 months after surgery. Corneal epithelial thickness and the Anterior stroma morphology were analyzed by using the NAVIS software V. 3.5.0 (NIDEK, Multi-Instrument Diagnostic System, Japan).

ELIGIBILITY:
Inclusion Criteria:

* Patients ask for PRK surgery
* Patients with stable refraction in the last year
* Patients without systemic and ocular disease
* Patients with 500 microns in pachymetry normal topography

Exclusion Criteria:

* Patients cannot attend their appointments
* Residual, recurrent or active ocular disease
* Previous ocular surgery except PRK
* Autoimmune or connective tissue disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-01; Primary Completion 2007-01 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
A central scan of the anterior stroma was taken with the confocal microscope (Confoscan 4, Fortune Technologies, Italy) | Before surgery and 1 week, 1 month, 3 months, 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ramirez F Manuel, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociación Para Evitar la Ceguera en Mëxico, Hospital "Luis Sánchez Bulnes"., Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Midena E, Gambato C, Miotto S, Cortese M, Salvi R, Ghirlando A. Long-term effects on corneal keratocytes of mitomycin C during photorefractive keratectomy: a randomized contralateral eye confocal microscopy study. J Refract Surg. 2007 Nov;23(9 Suppl):S1011-4. doi: 10.3928/1081-597X-20071102-06. PMID 18046999
- [Background] Ghirlando A, Gambato C, Midena E. LASEK and photorefractive keratectomy for myopia: clinical and confocal microscopy comparison. J Refract Surg. 2007 Sep;23(7):694-702. doi: 10.3928/1081-597X-20070901-08. PMID 17912939
- [Background] Ying L, Xiao Z, Liuxueying Z, Yumei J. Clinical use of in vivo confocal microscopy through focusing in corneal refractive surgery. J Refract Surg. 2006 Nov;22(9 Suppl):S1041-6. doi: 10.3928/1081-597X-20061102-07. PMID 17444091